CLINICAL TRIAL: NCT07364071
Title: Strategic ENdocrine and Targeted Radiation therapY
Brief Title: Strategic Endocrine Therapy and Targeted Radiotherapy for Prostate Cancer
Acronym: SENTRY
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Lantheus (Unknown)
Responsible Party: Principal Investigator, Tyler Seibert, Radiation Oncologist, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 813314
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma
Keywords: Radiotherapy; Androgen deprivation therapy; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RT + ST-ADT (Experimental): Radiotherapy with short-term androgen deprivation therapy (6 months) plus, if indicated, an androgen receptor pathway inhibitor.
  Interventions: Radiation: Radiation therapy
- RT + LT-ADT (Active Comparator): Radiotherapy with long-term androgen deprivation therapy (18 months).
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiotherapy with short-term androgen deprivation therapy plus, if indicated, an androgen receptor pathway inhibitor.

SUMMARY:
The goal of this clinical trial is to study definitive external beam radiation therapy together with drugs called androgen deprivation therapy (ADT) in patients with prostate cancer. The investigators want to find out if these drugs work the same way if they are given for 6 months or for the usual 18 months in patients who receive also definitive external beam radiotherapy. The investigators will also learn about the safety of the treatments. The main questions the study aims to answer are:

Do patients who get radiation therapy plus 6 months of androgen deprivation therapy need other hormone therapy or develop castration resistance at a higher rate within 5 years, compared to patients who get radiation therapy plus 18 months of androgen deprivation therapy?

Participants will:

Be treated with definitive external beam radiation therapy and receive androgen deprivation therapy for 6 months or 18 months.

Have visits once every 3 months for checkups and tests for at least 5 years. The visits at 3 months, 1 year, and 5 years need to be done in person; all the other visits can be done in person or remotely (telehealth).

Keep a diary of the missed doses of the androgen deprivation therapy.

DETAILED DESCRIPTION:
Definitive radiation therapy combined with hormone therapy improves oncologic outcomes in patients with high-risk prostate cancer. However, hormone therapy has substantial toxicity, including metabolic and cardiovascular, and negatively impacts quality-of-life. Previous trials demonstrated that long-term hormone therapy lasting 18-36 months improved overall survival compared to short-term hormone therapy lasting only 4-6 months. However, long-term hormone therapy also extends the duration of treatment-related toxicity. There is great interest among patients and physicians to reduce the total treatment time. A trial studying shorter duration of hormone therapy is warranted for the following reasons.

First, the trials that established the benefits of long-term hormone therapy were conducted over 20 years ago. Since then, advances in staging imaging and image-guided biopsy techniques have led to major stage migration in prostate cancer that has improved the prognosis of patients with disease categorized as high risk but localized. Second, substantial improvements in radiotherapy techniques have made it possible to deliver higher, more ablative radiation doses to the tumor while sparing normal organs. Third, even recurrent disease after definitive radiotherapy can now be detected early and managed with advanced radiotherapy (stereotactic ablative radiotherapy) to delay a need for salvage hormone therapy. Fourth, recent randomized trials have demonstrated that combining conventional androgen-deprivation therapy - usually accomplished with a gonadotropin-releasing hormone agonist or antagonist - with an androgen receptor pathway inhibitor is safe and improves overall survival in advanced prostate cancer.

These advances suggest that modern radiotherapy combined with short-term androgen deprivation therapy - and an optional androgen receptor pathway inhibitor - may achieve outcomes comparable to radiotherapy with long-term androgen deprivation therapy. This strategy offers the potential to maintain tumor control, reduce treatment-related morbidity, and improve patient survivorship. This randomized trial will compare the efficacy and toxicity of this novel treatment approach against the current standard of care. The investigators hypothesize that the novel treatment approach will have excellent disease control - comparable to that achieved with traditional long term androgen deprivation therapy - while improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate.
2. High-risk localized prostate cancer, defined as ≥1 of the following (per National Comprehensive Cancer Network or D'Amico criteria):

   1. Prostate specific antigen ≥ 20 ng/mL
   2. Gleason score 8-10
   3. Clinical stage T3a or higher; imaging can be used to determine T stage if there is macroscopic (gross) extraprostatic extension or invasion of the seminal vesicles or other non-prostate organs
3. No evidence of distant metastasis, confirmed by:

   a. Prostate-specific membrane antigen positron emission tomography/computed tomography (PSMA PET/CT) or equivalent staging imaging
4. Planning to receive definitive external beam radiotherapy and hormone therapy as standard of care (on label or medically accepted) treatment
5. Eastern Cooperative Oncology Group performance status 0-1.
6. Age ≥ 18 years.
7. Willingness to use adequate contraception if sexually active and of reproductive potential
8. Ability to understand and willingness to sign informed consent.
9. Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

1. Evidence of metastatic disease, including nodal disease beyond the pelvis or distant metastases on imaging.
2. Clear evidence of regional nodal disease on conventional imaging.
3. Prior prostatectomy.
4. Prior systemic therapy for prostate cancer, including:

   1. Androgen deprivation therapy (Note that participants who have started Androgen deprivation therapy within 90 days prior to randomization can be enrolled.)
   2. Androgen receptor pathway inhibitor (e.g., abiraterone, enzalutamide, apalutamide, darolutamide).
   3. Chemotherapy for prostate cancer.
5. Prior pelvic radiotherapy.
6. Any condition that, in the investigator's judgment, would compromise the patient's safety or compliance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients with prostate cancer can be enrolled.
Enrollment: 150 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | Within 5 years
  To compare failure-free survival of radiotherapy plus short-term androgen deprivation therapy plus, if indicated, an androgen receptor pathway inhibitor to that of radiotherapy plus long-term androgen deprivation therapy.
  Participants will be considered to have failure-free survival if they do not experience any of the events in the 5 years after the end of radiation therapy:
  1. Death from any cause.
  2. Initiation of salvage hormone therapy as defined in the protocol.
  3. Castration resistance per the Prostate Cancer Clinical Trials Working Group 3 definition. Castration resistance is defined as biochemical or clinical progression - as defined in the protocol - while serum testosterone is at castrate levels (<50 ng/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Seibert, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No